CLINICAL TRIAL: NCT05389124
Title: Functional Metagenomic Characterisation of Resilience in Experimental Gingivitis
Brief Title: Metagenome Resilience in Experimental Gingivitis
Status: Completed | Type: Observational
Sponsor: Newcastle University (Other)
Collaborators: Unilever SEAC (Industry); Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: NU008913
Record Dates: First submitted 2022-05-18; First posted 2022-05-25 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2022-05

CONDITIONS: Gingivitis; Oral Disease
Keywords: Experimental gingivitis; Dental plaque; Metagenome; Oral health
MeSH Terms: conditions — Gingivitis; Mouth Diseases; Dental Plaque

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gingival margin plaque.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental gingivitis: Group will wear a splint during oral hygiene to cover one quadrant of their dentition. They will develop gingivitis over 3 weeks. They will practise normal oral hygiene in the rest of their mouth (with minor restrictions, e.g. no mouthwash) and one other quadrant will act as an internal control for the gingivitis. After 3 weeks, normal oral hygiene will be restored throughout the mouth and subjects will continue to be monitored for a further 3 weeks.
  Interventions: Behavioral: Partial abstinence from oral hygiene

INTERVENTIONS:
Behavioral: Partial abstinence from oral hygiene — One quadrant of the dentition will be protected from oral hygiene for 3 weeks.

SUMMARY:
This study aims to identify new biomarkers that indicate the resilience of individuals to developing oral disease. An 'experimental gingivitis' model will be employed in which subjects will refrain from oral hygiene in one quadrant of their mouths for 3 weeks, and will then restore oral hygiene. Gum inflammation will be monitored by clinical measures throughout the trial and samples will be collected for analysis of microbial DNA and RNA.

DETAILED DESCRIPTION:
This project will employ an extended experimental gingivitis model to monitor changes in the oral metagenome and metatranscriptome during progression to gingivitis and recovery to oral health. The study will employ a 'split-mouth' design whereby one half of each individual's mouth is protected from oral hygiene while the other half acts as an internal control. Oral health status will be monitored through clinical measurements of dental plaque accumulation and gingival index. Plaque samples will be collected for DNA (metagenome) and RNA (metatranscriptome) sequencing. Using statistical modelling, genes and functional pathways will be identified that associate with resistance and resilience to gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* have read, understood and signed an informed consent form
* be adults of age 18 years or over
* have a minimum of 20 natural teeth (excluding third molars)
* be willing and able to comply with study procedures
* be a non-smoker and non-user of e-cigarettes or other oral intake nicotine replacement therapy (or have quit smoking/e-cigarettes/oral intake nicotine replacement therapy at least 2 years previously)
* healthy participants: good oral (no sites with interproximal attachment loss, GI ≥ 2.0 in ≤ 10% sites, %BOP scores ≤ 10%) and good general health.
* Covid-19 negative by LFT and fully vaccinated

Exclusion Criteria:

* infectious or systemic diseases that may be unduly affected by participation in this study
* extensive crown or bridge work and/or rampant decay at the discretion of the examiner
* wear removable partial dentures, a fixed/removable orthodontic appliance
* diabetes
* history of xerostomia, salivary gland disease, head and neck radiotherapy, Sjögren's syndrome, mucocutaneous disorders of the oral cavity, vesicobullous disorders of the oral cavity
* smoking or use of e-cigarettes within the last 2 years
* current use of prescription or over-the-counter medications that could affect salivary flow, at the discretion of the examiner
* lack of capacity to be able to consent to the research project and/or inability to follow study instructions
* pregnant by medical history or nursing
* currently undergoing or requiring extensive dental, orthodontic or implant treatment, or treatment for peri-implantitis
* treatment with antibiotics for any medical or dental condition within 4 weeks prior to enrolment
* scale and polish within 4 weeks prior to enrolment
* long term use of antibiotics or non-steroidal anti-inflammatory drugs (prophylactic low dose aspirin is permitted though)
* evidence of drug induced gingival overgrowth
* participation in a dental research study within the previous 20 days.
* Unilever personnel and personnel in the University department performing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gingivally healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Metagenomic sequence | Intervals up to 6 weeks
  Change from baseline

SECONDARY OUTCOMES:
Metatranscriptomic sequence | Intervals up to 6 weeks
  Change from baseline
Lobene Modified Gingival Index: Min 0 - Max 4; Worse- higher score indicates more gingival inflammation | Intervals up to 6 weeks
  Change from baseline
Plaque Index (Modified Quigley & Hein): Min 0 - Max 5; Worse - higher score indicates more plaque | Intervals up to 6 weeks
  Change from baseline
Bleeding Index (Bleeding on probing): Min 0 - Max 1; Worse- higher score indicates a bleeding site | Intervals up to 6 weeks
  Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Jakubovics, PhD, Study Director — Newcastle University; Richard Holliday, PhD, Principal Investigator — Newcastle University
Locations (1):
- Dental Clinical Research Facility, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised participant demographics will be linked to the data: Year of birth, sex, ethnicity.